CLINICAL TRIAL: NCT06418958
Title: In Vivo Temperature Changes Caused by Exposure to Short- and Long-wavelengths
Brief Title: Temperature Rise Caused by Short or Long-wavelengths
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB202300690; 1K23DE034470-01 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blue Light (Active Comparator): Light-curing procedure performed using blue light emission.
  Interventions: Device: Blue Light
- Red Light (Experimental): Light-curing procedure performed using red light emission.
  Interventions: Device: Red Light

INTERVENTIONS:
Device: Red Light — Light Curing with Red Light
  Arms: Red Light
Device: Blue Light — Light Curing with Blue Light
  Arms: Blue Light

SUMMARY:
Red light has been shown to be less harmful than blue light in vitro and in vivo. Although red light has been already introduced in the market and is currently being used in patients for several reasons, no data exist on the use of red light applied to restorative procedures. This study aims to specifically measure the in vivo temperature rise in simulated restorative procedures using blue light (standard) and red light and its post-operative sensitivity rates.

DETAILED DESCRIPTION:
Light-cured materials revolutionized dentistry as they allowed to control the setting of the materials in a timely manner simply upon light exposure. Although blue light has been routinely used to cure dental restorative materials for over 50 years, there are still potential risks to dental patients. These risks include gingiva burn or recession and pulp inflammation that can lead to necrosis in more severe situations due to the heat generated by this short wavelength (blue light). In addition, blue light has direct deleterious effects on cells, including irreversible imbalance in reactive oxygen species (ROS), damage to the mitochondrial DNA, and promoting collagen degradation. On the other hand, long wavelengths (such as red light) are known to have opposite effects, reducing inflammation and increasing cell proliferation. Although red light has been already introduced in the market and is currently being used in patients for several reasons, no in vivo data exist on the use of red-light applied to restorative procedures. Thus, this study aims to specifically measure the in vivo temperature rise in the tooth and gingival tissues surrounding restorative procedures using blue light (standard of care) and red light (investigational device) and evaluate/compare its post-operative sensitivity rates. The research hypothesis is that red light will generate less heat and less post-operative sensitivity than blue light (standard of care) while being used in dental restorative procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA I classification
* Fully erupted pre-molar(s);
* Absence of caries;
* Absence of restoration.

Exclusion Criteria:

* Radiographic constriction of the pulp chamber;
* Absence of apical closure;
* Formation of pulp stones or diffuse calcification at the pulp chamber;
* Presence of active carious lesions;
* Diagnosed reversible or irreversible pulpitis;
* Existing periapical lesion;
* Existing or planned root canal treatment.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Temperature Change | During restorative procedure.
  Temperature changes in degrees Celsius will be live-recorded by means of temperature probes for surface temperature acquisition.

SECONDARY OUTCOMES:
Post-Operative Sensitivity | One week (±2 days) after intervention.
  All patients will be called after the restoration(s) were placed to follow-up on any possible post-operative sensitivity or other questions or concerns. Post-operative sensitivity will be recorded as present or absent. If present, the post-operative sensitivity will be classified as mild, moderate, or severe according to the visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida College of Dentistry Dental Clinical Research Unit, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No